CLINICAL TRIAL: NCT00502541
Title: A Multicenter, Randomized, Masked, Controlled Study to Evaluate Retisert, and Intravitreal Fluocinolone Acetonide Implant, in the Treatment of Patients With Diabetic Macular Edema
Brief Title: Efficacy of Fluocinolone Acetonide Intravitreal Implant in Diabetic Macular Edema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDS FL-005; NCT00031525 (obsolete NCT alias)
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluocinolone acetonide (Experimental): Fluocinolone acetonide intravitreal implant
  Interventions: Drug: fluocinolone acetonide
- Standard of Care (Active Comparator): Standard of care
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: fluocinolone acetonide — fluocinolone acetonide 0.59 mg intravitreal implant
  Arms: Fluocinolone acetonide
Procedure: Standard of Care — Repeat macular grid laser or observation
  Arms: Standard of Care

SUMMARY:
This was a multi-center, randomized, masked, parallel-group, controlled study in patients with diabetic macular edema, comparing RetisertTM (0.59 mg) with control therapy (standard of care (SOC) - repeat macular grid laser or observation). The objective was to evaluate the safety and efficacy of the intravitreal fluocinolone acetonide implant in the treatment of patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant females at least 18 years of age, with DME in the study eye
* Edema must involve fixation and be at least 1 disc area in size
* Visual acuity of ≥20 and ≤68 letters by ETDRS in the study eye
* The study eye must have received at least one macular laser treatment > 12 weeks prior to entry into the study
* Ability and willingness to comply with treatment and follow-up
* Ability to understand and sign the Informed Consent form

Exclusion Criteria:

* Pregnant, lactating females
* Allergy to fluocinolone acetonide or any component of the delivery system
* Any disease or condition that would preclude study treatment or follow up
* Presence at screening of IOP greater or equal to 22 mm HG while on antiglaucoma medication(s).
* History of uncontrolled IOP within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2001-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
A change from baseline in visual acuity using ETDRS charts • Humphrey Visual Field Mean Defect (24-2) • Masked reading of the size of the area of retinal thickening on color photographs and OCT, where available, and of severity of fluorescein leakage | at 26 weeks and yearly through completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Background] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128